CLINICAL TRIAL: NCT06423703
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled Study to Evaluate the Efficacy and Safety of Cebranopadol for the Treatment of Moderate to Severe Acute Pain After Primary Unilateral Bunionectomy
Brief Title: A Study of Cebranopadol for the Treatment of Acute Pain After Bunionectomy
Acronym: ALLEVIATE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRN-228-302
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Pain
Keywords: Bunionectomy
MeSH Terms: conditions — Acute Pain | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cebranopadol (Experimental): once daily for 3 days
  Interventions: Drug: Cebranopadol; Drug: Placebo
- Oxycodone IR (Active Comparator): four times per day for 3 days
  Interventions: Drug: Oxycodone IR
- Placebo (Placebo Comparator): four times per day for 3 days
  Interventions: Drug: Placebo Only

INTERVENTIONS:
Drug: Cebranopadol — once daily for 3 days
  Other Names: TRN-228
  Arms: Cebranopadol
Drug: Oxycodone IR — four times per day for 3 days
  Other Names: oxycodone immediate release
  Arms: Oxycodone IR
Drug: Placebo Only — four times per day for 3 days
  Arms: Placebo
Drug: Placebo — three times per day for 3 days
  Arms: Cebranopadol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Cebranopadol for acute pain after a bunionectomy.

DETAILED DESCRIPTION:
This study is a Phase 3, multicenter, randomized, double-blind, placebo- and active-controlled parallel-group study to evaluate the efficacy and safety of cebranopadol in the treatment of postoperative pain following primary unilateral bunionectomy with first metatarsal osteotomy. The study will be conducted in 3 phases: Screening, Treatment, and Follow-up.

ELIGIBILITY:
Key Inclusion Criteria Before Surgery:

* Scheduled to undergo primary unilateral bunionectomy with first metatarsal osteotomy and internal fixation with no collateral procedures, using anesthesiologic and surgical procedures planned.
* Must be able to adhere to the visit schedule, complete all study assessments and protocol requirements, including self-reported questionnaires.

Key Exclusion Criteria Before Surgery:

* Any clinically significant disease, medical condition, or laboratory finding that in the investigator's opinion may interfere with the study procedures or data integrity, or compromise the safety of the subject.
* Secondary (i.e., unrelated to bunion) current painful condition that could confound the interpretation of efficacy, safety, or tolerability data in the study, in the opinion of the investigator.
* Subjects who require any analgesic for secondary (i.e., unrelated to bunion) painful condition that might impact the subject's ability to properly assess their postoperative pain, or that may require treatment during the Treatment Phase.
* History of allergy or hypersensitivity to any opioid analgesics, anesthetics, ibuprofen, or other NSAIDs.

Immediate Postoperative Exclusion Criteria:

* Surgical, postsurgical, or anesthetic complication that could confound the interpretation of efficacy, safety, or tolerability data in the study.
* Deviation from the surgical, postsurgical, or anesthetic protocol that could confound the interpretation of efficacy, safety, or tolerability data in the study.
* Evidence of hemodynamic instability or respiratory insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Pain NRS area under the curve: cebranopadol vs. placebo | 2-48 hours

SECONDARY OUTCOMES:
Proportion of subjects who require opioid rescue medication | 1-7 Days
Global Assessment of Satisfaction | 1-7 Days
Total oxycodone rescue consumption | 1-7 Days

OTHER OUTCOMES:
Incidence of Respiratory Safety Events | 1-7 Days

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Bertoch, MD, Principal Investigator — Cenexel JBR
Locations (10):
- United States (10):
  - ALLEVIATE 2 Site 001108, Sheffield, Alabama
  - ALLEVIATE 2 Site 001106, Little Rock, Arkansas
  - ALLEVIATE 2 Site 001103, Tampa, Florida
  - ALLEVIATE 2 Site 001102, Atlanta, Georgia
  - ALLEVIATE 2 Site 001107, Overland Park, Kansas
  - ALLEVIATE 2 Site 001105, Pasadena, Maryland
  - Alleviate 2 001113, Houston, Texas
  - ALLEVIATE 2 Site 001104, McAllen, Texas
  - ALLEVIATE 2 Site 001111, San Antonio, Texas
  - ALLEVIATE 2 Site 001101, Salt Lake City, Utah